CLINICAL TRIAL: NCT00799461
Title: INSPIRE: An Internet-based RCT for Long-term Survivors of Hematopoietic Stem Cell Transplantation
Brief Title: Internet-Based Program With or Without Telephone-Based Problem-Solving Training in Helping Long-Term Survivors of Hematopoietic Stem Cell Transplant Cope With Late Complications
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Syrjala, Karen, Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Organization: Fred Hutchinson Cancer Center (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2258.00; NCI-2009-01545 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); R01CA112631 (NIH)
Record Dates: First submitted 2008-11-26; First posted 2008-11-27 (Estimated); Last update posted 2012-03-07 (Estimated); Status verified 2012-03

CONDITIONS: Accelerated Phase Chronic Myelogenous Leukemia; Adult Acute Lymphoblastic Leukemia in Remission; Adult Acute Myeloid Leukemia in Remission; Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Atypical Chronic Myeloid Leukemia, BCR-ABL Negative; Blastic Phase Chronic Myelogenous Leukemia; Cancer Survivor; Chronic Eosinophilic Leukemia; Chronic Myelomonocytic Leukemia; Chronic Neutrophilic Leukemia; Chronic Phase Chronic Myelogenous Leukemia; de Novo Myelodysplastic Syndromes; Depression; Disseminated Neuroblastoma; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Fatigue; Long-term Effects Secondary to Cancer Therapy in Adults; Myelodysplastic/Myeloproliferative Neoplasm, Unclassifiable; Nodal Marginal Zone B-cell Lymphoma; Noncontiguous Stage II Adult Burkitt Lymphoma; Noncontiguous Stage II Adult Diffuse Large Cell Lymphoma; Noncontiguous Stage II Adult Diffuse Mixed Cell Lymphoma; Noncontiguous Stage II Adult Diffuse Small Cleaved Cell Lymphoma; Noncontiguous Stage II Adult Immunoblastic Large Cell Lymphoma; Noncontiguous Stage II Adult Lymphoblastic Lymphoma; Noncontiguous Stage II Grade 1 Follicular Lymphoma; Noncontiguous Stage II Grade 2 Follicular Lymphoma; Noncontiguous Stage II Grade 3 Follicular Lymphoma; Noncontiguous Stage II Mantle Cell Lymphoma; Noncontiguous Stage II Marginal Zone Lymphoma; Noncontiguous Stage II Small Lymphocytic Lymphoma; Previously Treated Myelodysplastic Syndromes; Primary Myelofibrosis; Psychosocial Effects of Cancer and Its Treatment; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Acute Myeloid Leukemia; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Hodgkin Lymphoma; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Cutaneous T-cell Non-Hodgkin Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Small Lymphocytic Lymphoma; Refractory Chronic Lymphocytic Leukemia; Refractory Hairy Cell Leukemia; Refractory Multiple Myeloma; Relapsing Chronic Myelogenous Leukemia; Secondary Acute Myeloid Leukemia; Secondary Myelodysplastic Syndromes; Splenic Marginal Zone Lymphoma; Stage I Multiple Myeloma; Stage II Multiple Myeloma; Stage III Adult Burkitt Lymphoma; Stage III Adult Diffuse Large Cell Lymphoma; Stage III Adult Diffuse Mixed Cell Lymphoma; Stage III Adult Diffuse Small Cleaved Cell Lymphoma; Stage III Adult Hodgkin Lymphoma; Stage III Adult Immunoblastic Large Cell Lymphoma; Stage III Adult Lymphoblastic Lymphoma; Stage III Chronic Lymphocytic Leukemia; Stage III Grade 1 Follicular Lymphoma; Stage III Grade 2 Follicular Lymphoma; Stage III Grade 3 Follicular Lymphoma; Stage III Mantle Cell Lymphoma; Stage III Marginal Zone Lymphoma; Stage III Multiple Myeloma; Stage III Small Lymphocytic Lymphoma; Stage IV Adult Burkitt Lymphoma; Stage IV Adult Diffuse Large Cell Lymphoma; Stage IV Adult Diffuse Mixed Cell Lymphoma; Stage IV Adult Diffuse Small Cleaved Cell Lymphoma; Stage IV Adult Hodgkin Lymphoma; Stage IV Adult Immunoblastic Large Cell Lymphoma; Stage IV Adult Lymphoblastic Lymphoma; Stage IV Chronic Lymphocytic Leukemia; Stage IV Grade 1 Follicular Lymphoma; Stage IV Grade 2 Follicular Lymphoma; Stage IV Grade 3 Follicular Lymphoma; Stage IV Mantle Cell Lymphoma; Stage IV Marginal Zone Lymphoma; Stage IV Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Myeloid, Accelerated Phase; Congenital Abnormalities; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Blast Crisis; Pdgfra-Associated Chronic Eosinophilic Leukemia; Leukemia, Myelomonocytic, Chronic; Leukemia, Neutrophilic, Chronic; Leukemia, Myeloid, Chronic-Phase; Depression; Fatigue; Myeloproliferative Disorders; Lymphoma, B-Cell, Marginal Zone; Primary Myelofibrosis; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Hairy Cell; Multiple Myeloma | interventions — Psychiatric Rehabilitation; Therapeutics; Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm I (full website access w/ PST; first study only) (Experimental): Patients receive full access to INSPIRE website for 6 months, which offers an individually tailored greeting home page with links to information on each of the target areas identified as being elevated on baseline assessment and how to manage the complications; a bulletin board with input from other survivors that is solicited, edited, and posted weekly; resource pages; and an opportunity to send secure messages with questions or comments. Patients also undergo 4-8 phone-based PST sessions with a behavioral health specialist.
  Interventions: Other: internet-based intervention; Other: questionnaire administration; Procedure: psychosocial assessment and care; Procedure: assessment of therapy complications; Procedure: management of therapy complications; Procedure: fatigue assessment and management; Other: counseling intervention
- Arm II (full website access without PST) (Experimental): Patients receive full access to INSPIRE website for 6 months as in arm I.
  Interventions: Other: internet-based intervention; Other: questionnaire administration; Procedure: psychosocial assessment and care; Procedure: assessment of therapy complications; Procedure: management of therapy complications; Procedure: fatigue assessment and management
- Arm III (delayed website access) (Sham Comparator): Patients do not have access to INSPIRE website for 6 months. After 6 months, patients receive full access to INSPIRE website for 3 months.
  Interventions: Other: internet-based intervention; Other: questionnaire administration; Procedure: psychosocial assessment and care; Procedure: assessment of therapy complications; Procedure: management of therapy complications; Procedure: fatigue assessment and management

INTERVENTIONS:
Other: internet-based intervention — Delayed access to online educational information and resources for managing long term complications of hematopoietic cell transplantation
Other: questionnaire administration — Completion of questions in an online format
Procedure: psychosocial assessment and care — Assessment and care of psychosocial aspects
  Other Names: psychosocial assessment; psychosocial assessment/care; psychosocial care; psychosocial care/assessment; psychosocial studies
Procedure: assessment of therapy complications — Evaluation of complications of treatment
Procedure: management of therapy complications — Managing therapy complications
  Other Names: complications of therapy, management of
Procedure: fatigue assessment and management — Assessing and managing fatigue
  Other Names: fatigue assessment/management
Other: counseling intervention — Counseling provided via telephone
  Other Names: counseling and communications studies
  Arms: Arm I (full website access w/ PST; first study only)

SUMMARY:
RATIONALE: A personalized Internet-based program may help improve fatigue, depression, and quality of life in long-term survivors of stem cell transplant. It is not yet known whether an Internet-based program is more effective with or without telephone-based problem-solving training.

PURPOSE: This randomized clinical trial is studying how well an Internet-based program works with or without telephone-based problem-solving training in helping long-term survivors of hematopoietic stem cell transplant cope with late complications

DETAILED DESCRIPTION:
OBJECTIVES:

I. To determine the efficacy of a randomized controlled trial to improve long term fatigue/physical dysfunction, depression/distress and health surveillance behaviors in adult 3 to 25-year hematopoietic stem cell transplant (HSCT) survivors using an internet only or internet and phone-based problem-solving and activation training compared with survivors randomized to a delayed internet access control.

II. To determine the reach, utilization, and implementation costs of a web-based, individually tailored intervention, disseminated through widely used patient information websites, targeting a national cohort of adult 2-25 year HSCT survivors. (Phase III/IV) III. To determine, in a randomized controlled trial, the efficacy of a nationally disseminated, internet-based, individually tailored intervention to improve long-term fatigue, distress and health promotion behaviors in HSCT survivors, compared with survivors randomized to a delayed internet access control. (Phase III/IV)

OUTLINE: Patients with elevated fatigue, depression, and/or distress at baseline are randomized to 1 of 3 arms (ARMS I, II, or III). Patients without elevated fatigue, depression or distress at baseline are randomized to 1 of 2 arms (ARMS II or III).

ARM I (FULL WEBSITE ACCESS WITH PROBLEM-SOLVING TRAINING [PST]; FIRST STUDY ONLY; CLOSED TO ACCRUAL): Patients receive full access to INSPIRE website for 6 months, which offers an individually tailored greeting home page with links to information on each of the target areas identified as being elevated on baseline assessment and how to manage the complications; a bulletin board with input from other survivors that is solicited, edited, and posted weekly; resource pages; and an opportunity to send secure messages with questions or comments. Patients also undergo 4-8 phone-based PST sessions with a behavioral health specialist.

ARM II (FULL WEBSITE ACCESS WITHOUT PST): Patients receive full access to INSPIRE website for 6 months as in ARM I.

ARM III (DELAYED WEBSITE ACCESS): Patients do not have access to INSPIRE website for 6 months. After 6 months, patients receive full access to INSPIRE website for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Hematopoietic stem cell transplant recipient between 3-25 years since last transplant
* Hematopoietic stem cell transplant recipient > = 2 years since last transplant (second, phase III/IV study only)
* Any type of transplant (autologous, allogeneic, myeloablative, non-myeloablative, marrow or peripheral blood stem cells)
* Able to communicate in English as indicated by ability to communicate adequately with study staff to participate in the clinical phone calls and to complete patient-reported outcomes (PRO) assessments in English
* Has internet and email access (indicated by logon to site for consent and assessment)

Exclusion Criteria:

* Does not complete the baseline assessment through the HADS (Hospital Anxiety and Depression Scale)
* Does not complete required assessments in the background and medical history forms required to determine whether meet inclusion and exclusion criteria, stratification, sample description, or primary outcomes (includes age, gender, ethnicity, race, transplant site, and medical information about transplant if not FHCRC or SCCA patient, education, work, height and weight, current medications
* Survivors who score 3.0 or above on the SCL depression measure (indicating severe depression) or who report moderate to severe suicidal ideation will be ineligible for randomization; these survivors will, however, have full access to the website if they have completed the required baseline assessment; they will be asked to also complete follow-up assessments
* Survivors who report to us that they have been in active treatment for relapse of their original disease, or for a second cancer, in the past 2 years will be ineligible for randomization, unless the second cancer was treated only with surgical removal (e.g., basal, squamous or localized melanoma skin cancer, or breast ductal carcinoma in situ [DCIS])
* These survivors will, however, have full access to the website if they have completed the required baseline assessment; they will be asked to also complete follow-up assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1337 (Actual)
Dates: Start 2008-08; Primary Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Aggregate number of targeted problems | At 6 months
Reach of web-based intervention (second, phase III/IV study only) | At 6 months
  As indicated by proportion logging on the website content for males (targeting 50%), older (targeting 50% over age 55), and geographically underserved participants (targeting 20% rural residents as indicated by zip code), as well as percent who logon to the study website content after initially registering for the study (targeting 90%) second
Utilization of web-based intervention (second, phase III/IV study only) | At 6 months
  As indicated by number of pages viewed (targeting a mean of 10), log-on times (targeting a mean of 2) and time from notification of website content access to website content logon (targeting a mean of 2 weeks)
Satisfaction, use and barriers ratings at the end of the study including barriers to website use and barriers to using health promotion guidelines (second, phase III/IV study only) | At 6 months
Cost to maintain the site content (not including costs for maintenance of the assessment process) (second, phase III/IV study only) | At 6 months
  As indicated by per participant prorated costs for materials and time for updating content, responding to participant comments and requests, maintaining programming and responding to technical problems

SECONDARY OUTCOMES:
Mean z score combining the Vitality and Physical Function subscales of the SF-36 | At 6 months
Mean z score combining the Symptom Checklist 90-R Depression scale and the Cancer and Treatment Distress - Uncertainty subscale | At 6 months
Total health care utilization behaviors | At 6 months
Long-term fatigue and distress of survivors compared with controls (second, phase III/IV study only) | At 6 months
Long-term health promotion of survivors compared with controls (second, phase III/IV study only) | At 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Karen Syrjala, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States

REFERENCES:
- [Derived] Walsh CA, Yi JC, Leisenring WM, Syrjala KL. Social Support, Coping, and Cancer-Related Health Burden in Long-term Survivors Treated with Hematopoietic Stem Cell Transplantation as Adolescents or Young Adults. J Adolesc Young Adult Oncol. 2023 Aug;12(4):496-502. doi: 10.1089/jayao.2022.0105. Epub 2022 Oct 25. PMID 36282798
- [Derived] Norskov KH, Yi JC, Crouch ML, Fiscalini AS, Flowers MED, Syrjala KL. Social support as a moderator of healthcare adherence and distress in long-term hematopoietic cell transplantation survivors. J Cancer Surviv. 2021 Dec;15(6):866-875. doi: 10.1007/s11764-020-00979-4. Epub 2021 Jan 9. PMID 33420905
- [Derived] Walsh CA, Yi JC, Rosenberg AR, Crouch MV, Leisenring WM, Syrjala KL. Factors associated with social functioning among long-term cancer survivors treated with hematopoietic stem cell transplantation as adolescents or young adults. Psychooncology. 2020 Oct;29(10):1579-1586. doi: 10.1002/pon.5460. Epub 2020 Aug 13. PMID 32628342